CLINICAL TRIAL: NCT02445703
Title: Phase IV Immunogenicity and Safety Study of Different Immunization Schedules of Inactivated Hepatitis A Vaccine (HAV) and/ or Combined Hepatitis A and Hepatitis B Vaccine (HABV) in Healthy Chinese Infants
Brief Title: Comparison of Immunization Schedules of Inactivated Hepatitis A Vaccine and Combined Hepatitis A and Hepatitis B Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-HAB-4005
Record Dates: First submitted 2015-05-13; First posted 2015-05-15 (Estimated); Last update posted 2021-07-27 (Actual); Status verified 2015-05

CONDITIONS: Hepatitis A; Hepatitis B
MeSH Terms: conditions — Hepatitis A; Hepatitis B | interventions — Hepatitis B Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (HAV + HAV) (Experimental): Intervention: Inactivated Hepatitis A vaccine (HAV);
  Subjects in this group each received 2 doses of inactivated HAV with a 6-month interval (day 0, month 6);
  Route of administration: intramuscular injection in deltoid region;
  Interventions: Biological: Inactivated Hepatitis A vaccine (HAV)
- Group 2 (HAV + HABV) (Experimental): Intervention: Inactivated Hepatitis A vaccine (HAV) and Combined hepatitis A and hepatitis B vaccine (HABV);
  Subjects in this group each received 1 dose of inactivated HAV at day 0, and 1 dose of HABV at month 6.
  Route of administration: intramuscular injection in deltoid region;
  Interventions: Biological: Inactivated Hepatitis A vaccine (HAV); Biological: Combined hepatitis A and hepatitis B vaccine (HABV)
- Group 3 (HABV + HABV) (Experimental): Intervention: Combined hepatitis A and hepatitis B vaccine (HABV);
  Subjects in this group each received 2 doses of HABV with a 6-month interval (day 0, month 6);
  Route of administration: intramuscular injection in deltoid region;
  Interventions: Biological: Combined hepatitis A and hepatitis B vaccine (HABV)

INTERVENTIONS:
Biological: Inactivated Hepatitis A vaccine (HAV) — Dosage of HAV is 250u hepatitis A antigen/0.5ml/dose.
  Other Names: Healive (Sinovac Biotech Ltd.); lot No.: 201308046
  Arms: Group 1 (HAV + HAV); Group 2 (HAV + HABV)
Biological: Combined hepatitis A and hepatitis B vaccine (HABV) — Dosage of HABV is 250u hepatitis A antigen and 5µg hepatitis B antigen/0.5ml/dose
  Other Names: Bilive (Sinovac Biotech Ltd.); lot No.: 201307017
  Arms: Group 2 (HAV + HABV); Group 3 (HABV + HABV)

SUMMARY:
The purpose of this study is to compare the immunogenicity and safety of three different immunization schedules of inactivated hepatitis A vaccine (HAV) and/ or combined hepatitis A and B vaccine (HABV) in healthy Chinese infants.

DETAILED DESCRIPTION:
This study is a randomized double-blind, single-center, phase IV clinical trial. The purpose of this study is to compare the immunogenicity and safety of three different immunization schedules of inactivated hepatitis A vaccine (HAV) and/ or combined hepatitis A and B vaccine (HABV) in healthy Chinese infants between 18 and 24 months old. The subjects were randomly assigned into 3 groups. Subjects in group 1 each received 2 doses of HAV with a 6-month interval (at day 0 and month 6); subjects in group 2 each received 1 dose of HAV at day 0 and 1 dose of HABV at month 6; subjects in group 3 each received 2 doses of HABV with a 6-month interval (at day 0 and month 6).

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants between 18 and 24 months old;
* Have not received hepatitis A vaccine before;
* Completed hepatitis B vaccine full immunization schedule;
* Written consent of the guardian of each participant;

Exclusion Criteria of the First Injection:

* History of allergy to vaccine(s), or history of serious adverse reaction to vaccination, such as urticaria, dyspnea, angioneurotic edema, or abdominal pain;
* Autoimmune disease or immunodeficiency;
* Any acute disease that made the conditions of the person unsuitable for vaccination
* Administration of any live attenuated vaccine within 14 days prior to the injection;
* Administration of any subunit vaccine or inactivated vaccine within 7 days prior to the injection;
* Administration of treatment of immunosuppressants (e.g., corticosteroid) within 1 month prior to the injection, or planning for such treatment during this study;
* Body temperature > 37.0 °C before injection;
* Based on the evaluation of the investigator, there was any other factor that indicating the person was unsuitable for this study;

Exclusion Criteria of the Second Injection:

* Any acute infectious disease, body temperature > 38.5 °C or acute attacks of chronic diseases within 3 days prior to the second injection;
* Administration of blood product or other investigational drug during this study;
* Occurrence of adverse event at grade 3 or higher and the event was related to the first injection;
* The investigator or the Ethic Committee decided that the subject should be excluded;

Ages: 18 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 301 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The Post-immunization Seropositivity Rates (SPR) to Hepatitis A | 7 months
  The post-immunization SPR is the percent of participants with anti-HAV titers ≥ 20 mIU/mL at month 7. Anti-HAV titers were detected in participants' serum samples using electrochemiluminescence immunoassay.

SECONDARY OUTCOMES:
The Post-immunization Geometric Mean Concentration (GMC) of Hepatitis A Antibody (anti-HAV) | 7 months
  The post-immunization GMC values of anti-HAV were measured using electrochemiluminescence immunoassay in serum samples collected at month 7.
The Post-immunization GMC of Hepatitis B Surface Antibody (HBsAb) | 7 months
  The post-immunization GMC values of HBsAb were detected using electrochemiluminescence immunoassay in serum samples collected at month 7.
The Post-immunization SPR to Hepatitis B | 7 months
  The post-immunization SPR is the percent of participants with HBsAb titer ≥ 10 mIU/mL at month 7. HBsAb titers were detected in participants' serum samples using electrochemiluminescence immunoassay.
Occurrence of Adverse Events (AEs) | 7 months
  AE information was collected after first injection (day 0) until month 7. Each AE case was reviewed by the investigator to determine whether or not it was an adverse reaction (related to the vaccination). After each injection, a 30-minute safety observation was conducted immediately, and body temperature and solicited adverse events (AEs) within 72 hours were recorded. Unsolicited AEs information was collected from day 0 (after injection) to month 7.

CONTACTS AND LOCATIONS:
Overall Officials: Fangjun Li, BS, Principal Investigator — Hunan Provincial Center for Disease Control and Prevention
Locations (1):
- Hunan Provincial Center for Disease Control and Prevention, Changsha, Hunan, China

REFERENCES:
- [Derived] Li F, Hu Y, Zhou Y, Chen L, Xia W, Song Y, Tan Z, Gao L, Yang Z, Zeng G, Han X, Li J, Li J. A Randomized Controlled Trial to Evaluate a Potential Hepatitis B Booster Vaccination Strategy Using Combined Hepatitis A and B Vaccine. Pediatr Infect Dis J. 2017 May;36(5):e157-e161. doi: 10.1097/INF.0000000000001535. PMID 28060048